CLINICAL TRIAL: NCT04358588
Title: Expanded Access: Pulsed, Inhaled Nitric Oxide (iNO) for the Treatment of Patients With Mild or Moderate Coronavirus Disease (COVID-19)
Brief Title: Pulsed Inhaled Nitric Oxide for the Treatment of Patients With Mild or Moderate COVID-19
Status: No longer available | Type: Expanded Access
Sponsor: Bellerophon (Industry)
Responsible Party: Sponsor
Other Study IDs: PULSE-EAP-001
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus Infection; COVID-19; Pneumonia, Viral
Keywords: coronavirus; corona virus; COVID-19; COVID 19; SARS; SARS-coronavirus; Pneumonia; Pneumonia, viral; Virus
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Pneumonia, Viral; Severe Acute Respiratory Syndrome; Pneumonia; Virus Diseases | interventions — Inosine

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: iNO (inhaled nitric oxide) delivered via the INOpulse Delivery System — Patients will be treated by means of an INOpulse device and cannula. The active study drug, nitric oxide for inhalation (iNO), will be provided in size 0.074 liter aluminum cartridge at a concentration of 6.0 mg/L (4880 ppm).

SUMMARY:
The search for novel therapies to address the ongoing coronavirus (COVID-19) pandemic is ongoing. No proven therapies have been identified to prevent progression of the virus. Preliminary data suggest that inhaled nitric oxide (iNO) could have benefit in preventing viral progression and reducing reliance on supplemental oxygen and ventilator support.

Expanded access allows for iNO to be delivered via the portable INOpulse delivery system for the treatment of COVID-19.

DETAILED DESCRIPTION:
NO is a naturally produced molecule that is critical to the immune response to defend against pathogens and infections. In vitro studies have shown that NO inhibits the replication of severe acute respiratory syndrome-related coronavirus (SARS-CoV) and improves survival for cells infected with SARS-CoV. Additionally, in a clinical study of patients infected with SARS-CoV, iNO demonstrated improvements in arterial oxygenation, a reduction in ventilation support and an improvement in lung infiltrates observed on chest radiography. Based on the genetic similarities between the two coronaviruses, the data in SARS-CoV support the potential for iNO to provide meaningful benefit for patients infected with COVID-19.

The clinical spectrum of the COVID-19 infection ranges from mild signs of upper respiratory tract infection to severe pneumonia and death. Preventing disease progression in patients with mild or moderate disease would improve morbidity/mortality and significantly reduce the impact on limited healthcare resources.

Expanded access allows for iNO to be delivered via the INOpulse delivery system for the treatment of COVID-19. INOpulse technology provides targeted pulsatile delivery of iNO via portable INOpulse delivery system.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (and assent as appropriate) prior to the initiation of any study mandated procedures or assessments.
2. At least 18 years old
3. Patients with proven or high suspicion of SARS-CoV-2 infection and on supplemental oxygen ≤ 10 L/minute
4. Suspected or proven pneumonia on chest imaging
5. Female patients of childbearing potential must have a negative pre-treatment pregnancy test (serum or urine). All female patients should take adequate precaution to avoid pregnancy.
6. Willing and able to comply with treatment schedule and study procedures.

Exclusion Criteria:

1. Participating in any other clinical trial of an experimental treatment for COVID-19
2. Gas exchange and ventilation requiring the use of any continuous positive airway pressure (CPAP), or any system of Non Invasive Ventilation (NIV), with Positive End-Expiratory Pressure (PEEP) ≤ 10 cmH2O prior to initiation of iNO
3. Pregnancy, or positive pregnancy test in a pre-dose examination
4. Open tracheostomy
5. Clinical contra-indication, as deemed by the attending physician
6. Use of a nitric oxide donor agent such as nitroglycerin or drugs known to increase methemoglobin such as lidocaine, prilocaine, benzocaine or dapsone at screening
7. Known history or clinical evidence of heart failure, left ventricular dysfunction (LVEF < 40 %)
8. Patients reporting hemoptysis

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ashika Ahmed, MD, Study Director — Bellerophon Therapeutics

REFERENCES:
- [Background] Keyaerts E, Vijgen L, Chen L, Maes P, Hedenstierna G, Van Ranst M. Inhibition of SARS-coronavirus infection in vitro by S-nitroso-N-acetylpenicillamine, a nitric oxide donor compound. Int J Infect Dis. 2004 Jul;8(4):223-6. doi: 10.1016/j.ijid.2004.04.012. PMID 15234326
- [Background] Akerstrom S, Mousavi-Jazi M, Klingstrom J, Leijon M, Lundkvist A, Mirazimi A. Nitric oxide inhibits the replication cycle of severe acute respiratory syndrome coronavirus. J Virol. 2005 Feb;79(3):1966-9. doi: 10.1128/JVI.79.3.1966-1969.2005. PMID 15650225
- [Background] Chen L, Liu P, Gao H, Sun B, Chao D, Wang F, Zhu Y, Hedenstierna G, Wang CG. Inhalation of nitric oxide in the treatment of severe acute respiratory syndrome: a rescue trial in Beijing. Clin Infect Dis. 2004 Nov 15;39(10):1531-5. doi: 10.1086/425357. Epub 2004 Oct 22. PMID 15546092